CLINICAL TRIAL: NCT01455285
Title: Investigation of the Effectiveness of Different Modulations of Pulse Frequency Transcutaneous Electrical Nerve Stimulation in Dysmenorrhea
Brief Title: Effectiveness of the Transcutaneous Electrical Nerve Stimulation in Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Piauí (Other)
Purpose: Treatment
Other Study IDs: 0377.0.045.000-10
Record Dates: First submitted 2011-10-11; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-05

CONDITIONS: Dysmenorrhea
Keywords: dysmenorrhea; transcutaneous electrical nerve stimulation (TENS; analgesia; pain visual analog scale; McGill pain questionnaire
MeSH Terms: conditions — Dysmenorrhea; Agnosia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: transcutaneous electrical nerve stimulation

SUMMARY:
Hypothesis: What is the best modulation of pulse frequency in transcutaneous electrical nerve stimulation in dysmenorrhea? Purpose: To determine the effect of hypoalgesia frequency modulation pulse by transcutaneous electrical nerve (TENS) in dysmenorrhea. Methods: A controlled clinical study and prospective developed at the School of Physiotherapy Clinic / UFPI. Forty students were randomized into four distinct groups of the modulation frequency TENS: group 1 - 100 Hz, 100μs, group 2 - 4 Hz, 100μs, group 3 - placebo (apparatus off), group 4 - placebo induced (2 Hz, 40μs). All were initially evaluated by a questionnaire developed for the study, the visual analogue scale (VAS) (before, after 20, 30, 40, 50, 60 minutes) and the McGill Pain Questionnaire (before and after 20 minutes). The total duration of TENS application was 20 minutes and all protocols were performed in a single session. The analysis of variance (One-way ANOVA) followed by the Tukey procedure was applied to identify differences between experimental groups for each variable analyzed. The level of significance was p< 0,05.

ELIGIBILITY:
Inclusion Criteria:

* be the first or second day of menstruation
* dysmenorrhea present at the time of application of TENS
* not having undergone any procedure analgesic six hours before the application of TENS

Exclusion Criteria:

* not to mention dysmenorrhea at the time of evaluation
* pregnant women
* were using some method of hormonal contraception on an ongoing basis
* had sensory deficits or cognitive and cases of contraindication to TENS application.

Ages: 16 Years to 33 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physiotherapy Clinic UFPI / Campus Minister Reis Velloso, Parnaíba, Piauí, Brazil

REFERENCES:
- [Result] Proctor ML, Smith CA, Farquhar CM, Stones RW. Transcutaneous electrical nerve stimulation and acupuncture for primary dysmenorrhoea. Cochrane Database Syst Rev. 2002;2002(1):CD002123. doi: 10.1002/14651858.CD002123. PMID 11869624